CLINICAL TRIAL: NCT04339465
Title: Children Affected by Rare Disease and Their Families Network
Acronym: CARE-FAM-NET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silke Wiegand-Grefe, Prof. Dr. (Other)
Collaborators: Techniker Krankenkasse (Other); BARMER (Other); DAK Gesundheit (Other); KKH Kaufmännische Krankenkasse (Unknown); BKK Mobil Oil (Industry); Achse e.V. (Unknown); University of Ulm (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Schleswig-Holstein (Other); University Medical Center Rostock (Other); University Hospital Muenster (Other); University Hospital, Essen (Other); Ruhr University of Bochum (Other); Universitätsklinikum Köln (Other); University of Göttingen (Other); Hannover Medical School (Other); Evangelisches Klinikum Bethel (Unknown); Charite University, Berlin, Germany (Other); DRK Kliniken Berlin Westend (Unknown); Universitätsklinikum Leipzig (Other); University of Giessen (Other); University Hospital Freiburg (Other); Josefinum Augsburg (Unknown); University Hospital Augsburg (Other); University Hospital, Saarland (Other); Jena University Hospital (Other); Leibniz Universität, Center for Health Economics Research Hannover (Unknown); aQua-Institut (Unknown)
Responsible Party: Sponsor-Investigator, Silke Wiegand-Grefe, Prof. Dr., Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: U1111-1223-2871
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Rare Diseases
Keywords: rare disease; children and adolescents; e-mental health; early detection and early treatment of mental disorders
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized controlled multicenter study (RCT) with a factorial design with four groups: CAREFAM (face to face), WEP-CARE (online), both interventions, control group (TAU = treatment as usual).
Who Masked: Investigator
Masking Description: Assessors are blind regarding the randomization (group affiliation) of the families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CARE-FAM (Experimental): The face-to-face intervention CARE-FAM is a family-based intervention for the diagnostic, early detection and early treatment of mental health issues of children affected by rare diseases, their siblings and their parents. CARE-FAM is a brief low-frequency intervention comprising six to eight sessions per family over a period of six months. Following a preliminary talk, 2 sessions with the parents, 1 session with each affected child and each sibling and 3 sessions with the whole family will take place. This low-frequency approach (sessions every 2 to 3 weeks) allows families to integrate the intervention into their daily life. Upon request, the sessions will take place at the family's home (home-treatment).
  Interventions: Behavioral: CARE-FAM
- WEP-CARE (Experimental): The online intervention WEP-CARE addresses parents of children and adolescents affected by rare diseases. The program is based on principles of cognitive-behavioral writing therapy. Supported by trained professionals, the participants perform 12 standardized writing tasks on a secured internet platform. The 12 writing tasks will be conducted with a weekly frequency and participants will receive personalized feedback. WEP-CARE aims at enhancing mental health problems and the coping strategies of the family.
  Interventions: Behavioral: WEP-CARE
- CARE-FAM + WEP-CARE (Experimental): The families will receive both the face-to-face intervention CARE-FAM and the online intervention WEP-CARE.
  Interventions: Behavioral: CARE-FAM; Behavioral: WEP-CARE
- Treatment as usual (No Intervention): The treatment as usual implies that families of the control group receive the treatment that is customary in regular care. Thus, these families normally don't receive any post-treatment. If, however, a member of a control group family appears to have an urgent need for treatment (every family receives a comprehensive diagnostic investigation at the beginning of the study), the respective family will be placed in the ambulatory care system.

INTERVENTIONS:
Behavioral: CARE-FAM — CARE-FAM is a family-based intervention for the diagnostic, early detection and early treatment of mental health issues of children affected by rare diseases, their siblings and their parents. CARE-FAM is a brief low-frequency intervention comprising six to eight sessions per family over a period of six months.
  Arms: CARE-FAM; CARE-FAM + WEP-CARE
Behavioral: WEP-CARE — WEP-CARE is an online-intervention that addresses parents of children and adolescents affected by rare diseases. The program is based on principles of cognitive-behavioral writing therapy. Supported by trained professionals, the participants perform 12 standardized writing tasks on a secured internet platform
  Arms: CARE-FAM + WEP-CARE; WEP-CARE

SUMMARY:
Families of children with rare diseases (i.e., not more than 5 out of 10.000 people are affected) are often highly burdened with fears, insecurities and concerns regarding the affected child and his/her siblings. The project at hand will test two innovative forms of care (CARE-FAM and WEP-CARE) at 17 sites in 12 federal states of Germany. The goal is to improve the mental health and quality of life of children affected by rare diseases and their relatives in a sustainable manner. If successful, these interventions will be introduced into regular care.

DETAILED DESCRIPTION:
The central objective of the study at hand is to close the supply gap for families with children and adolescents affected by rare diseases. Two innovative forms of care (CARE-FAM and WEP-CARE) will be implemented and evaluated at the 18 participating study sites. Both interventions include psychological diagnostics, early detection and treatment of concomitant mental diseases. The study is a prospective, randomized controlled multicenter study (RCT) with a factorial design with four groups: CAREFAM (face to face), WEP-CARE (online), both interventions, control group (TAU = treatment as usual). Central psychosocial outcomes will be assessed at four time points (i.e., Baseline and after six, 12 and 18 months) from the perspectives of the parents, the affected child and the siblings (0 - 9 years only external assessment; from 10 years of age additional self-assessment) and the professionals.

ELIGIBILITY:
Inclusion Criteria:

1. Family with at least one child between 0 and 21 years with a rare disease or a suspected rare disease.
2. Consent to participate in the study.
3. Sufficient knowledge of the German language of parents and children.
4. Insured at the participating insurance companies.

Exclusion Criteria: Severe psychiatric disorders and impairments with acute symptoms such as suicidal tendencies, severe depression, addictions, acute psychotic symptoms etc., which will not be sufficiently supplied by this new low-frequency intervention. Children and parents with acute treatment demand in the control group will be placed at psychotherapists. Nevertheless, they stay in the control group.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 687 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mental health of parents (SCID) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Proportion of parents without mental abnormities among the parents with initial mental abnormities, assessed by the external, independent "Structured clinical interview for DSM-IV" (SCID; Wittchen, Zaudig & Fydrich,1997) 18 months after.

SECONDARY OUTCOMES:
Sociodemographic information of the parents | At baseline of the study
  Sociodemographic information of the parents, assessed from the perspective of the parents by ad-hoc items at the beginning of the study.
Health-related quality of life of the parents (EQ-5D) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the parents, assessed from the perspective of the parents by the EQ-5D (Brooks, Rabin & Charro, 2003; Hinz, Klaiberg, Brahler & Konig, 2006) at the beginning of the study as well as six, 12 and 18 months after the randomization.
Health-related quality of life of the parents (ULQIE) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the parents, assessed from the perspective of the parents by the "Ulmer Lebensqualitäts-inventar für Eltern chronisch kranker Kinder" (ULQIE; Goldbeck & Storck, 2002) at the beginning of the study as well as six, 12 and 18 months after the randomization.
Health-related quality of life of the parents (SF-12) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the parents, assessed from the perspective of the parents by the "Short Form 12" (SF-12; Bullinger & Kirchberger, 1998) at the beginning of the study as well as six, 12 and 18 months after the randomization.
Health-related quality of life of the chronically-ill children/adolescents (Kidscreen-27) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the chronically-ill children/adolescents and of the siblings, assessed from the perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the Kidscreen-27 (The KIDSCREEN Group Europe, 2006).
Health-related quality of life of the chronically-ill children/adolescents (DCGM-37) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Health-related quality of life of the chronically-ill children/adolescents, assessed from the perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the "Disabkids Chronic Generic Measure" (DCGM-37; Bullinger, Schmidt, Petersen & The DISABKIDS Group, 2002) at the beginning of the study as well as six, 12 and 18 months after the randomization.
Mental health of the parents (PHQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the parents, assessed from the perspective of the parents by the "Patient Health Questionnaire" (PHQ; Löwe, Spitzer, Zipfel & Herzog, 2002).
Mental health of the parents (BSI) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the parents, assessed from the perspective of the parents by the "Brief Symptom Inventory" (BSI; Franke, 2000).
Mental health of the chronically-ill children/adolescents and the siblings (Kiddie-SADS-PL) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Mental health of the chronically-ill children/adolescents and the siblings, assessed from the perspective of the parents and from the perspective of the children/adolescents (from 10 years of age) by an external independent interview "Diagnostic Interview Kiddie-Sads-Present and Lifetime Version" (Kiddie-SADS-PL; Delmo, Weiffenbach, Gabriel, Stadler & Poustka, 2001).
Psychiatric disorders of the chronically-ill children/adolescents and the siblings (CBCL) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Psychiatric disorders of the chronically-ill children/adolescents and the siblings, assessed from the perspective of the parents by the "Child Behaviour Checklist" (CBCL; Döpfner, Pflück, Kinnen & Arbeitsgruppe Deutsche Child Behavior Checklist, 2014).
Psychiatric disorders of the chronically-ill children/adolescents and the siblings (YSR) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Psychiatric disorders of the chronically-ill children/adolescents and the siblings, assessed from the perspective of the children/adolescents (from 10 years of age) by the "Youth Self Report" (YSR; Döpfner, Pflück, Kinnen & Arbeitsgruppe Deutsche Child Behavior Checklist, 2014).
Coping of the parents (CHIP-D) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Coping of the parents, assessed from the perspective of the parents by the German version of the "Coping Health Inventory for Parents" (CHIP-D; McCubbin, McCubbin, Cauble & Goldbeck, 2001).
Coping of the chronically-ill children/adolescents and the siblings (Kidcope) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Coping of the chronically-ill children/adolescents and the siblings, assessed from the perspective of the children/adolescents (from 10 years of age) by the "Kidcope Checklist" (Kidcope; Spirito, Stark & Williams, 1988).
Social support of the parents, of the chronically-ill children/adolescents and of the siblings (OSSQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Social support of the parents, of the chronically-ill children/adolescents and of the siblings, assessed from the perspective of the parents, of the chronically-ill children/adolescents and from the sibling, respectively, by the "Oslo Social Support Questionnaire" (OSSQ; Dalgard, 2006).
Family functioning (GARF) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Family functioning, assessed from the perspective of the therapist by the "Global Assessment of Relational Functioning" (GARF; Saß, Wittchen, Zaudig & Houben, 2003).
Relationships between siblings (SRQ) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Sibling relationship, assessed from the perspective of the siblings (from 10 years of age) by the "Sibling Relationship Questionnaire" (SRQ; Fuhrmann & Burmester, 1985).
Satisfaction with the relationship and parenting relationship of the parents (PFB) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Satisfaction with the relationship and parenting relationship of the parents, assessed from the perspective of the parents by the "Partnerschaftsfragebogen" (PFB; Hahlweg, 2016).
Eating behaviour of the chronically-ill children/adolescents (EDY-Q) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Eating behaviour of the chronically-ill children/adolescents, assessed from the perspective of the parents and from the perspective of the chronically-ill children/adolescents (from 10 years of age) by the "Eating Disorders in Youth - Questionnaire" (EDY-Q; van Dyck & Hilbert, 2016).
Body-related eating behaviour of the chronically-ill children/adolescents (ChEDE-Q8) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Body-related eating behaviour of the chronically-ill children/adolescents, assesse from the persepective of the chronically-ill children/adolescents (from 10 years of age) by the "Eating Disorder Examination - Questionnaire (Short Form)" (ChEDE-Q8; Kliem, Schmidt, Vogel, Hiemisch, Kiess & Hilbert, 2017).
Elimination disorders of the chronically-ill children/adolescents (Anamnesebogen Enuresis/Funktionelle Harninkontinenz) | Change from baseline of the study at 6,12 and 18 months after the randomization
  Elimination disorders of the chronically-ill children/adolescents, assessed from the perspective of the parents by the "Anamnesebogen Enuresis/Funktionelle Harninkontinenz" (von Gontard, 2010).
Treatment costs of the parents (CSSRI-DE) | Change from baseline of the study at 6 months after the randomization
  Treatment costs of the parents, assessed from the perspective of an external rater by the German version of the "Client Socioeconomic and Services Receipt Inventory" (CSSRI-DE; Roick, Kilian, Matschinger, Bernert, Mory & Angermeyer, 2001).
Treatment costs of the chronically-ill children/adolescents and the siblings (CAMHSRI-DE) | Change from baseline of the study at 6 months after the randomization
  Treatment costs of the chronically-ill children/adolescents and the siblings, assessed from the perspective of an external rater by the German version of the "Children and adolescent mental health services receipt inventory" (CAMHSRI-DE; Kilian, Losert, McDaid, Park, Knapp, Beecham, Kusakovskaja, Murauskiene & the CAMHEE Project, 2009).
Treatment assessment (FBB-T) | Change from 6 months after randomization at 12 and 18 months.
  Treatment assessment of the parents and the chronically ill children/adolescents and their siblings, in self-assessment from the age of 10 years and by the therapist, assessed on the basis of the treatment assessment questionnaire (FBB-T; Mattejat & Remschmid, 1998).
Patient satisfaction (ZUF-8) Patient satisfaction | Change from 6 months after randomization at 12 and 18 months.
  Patient satisfaction of the parents and the chronically ill children/adolescents and their siblings, assessed on the basis of the questionnaire on patient satisfaction (ZUF-8; Schmid & Nübling, 2002).

CONTACTS AND LOCATIONS:
Locations (17):
- Germany (17):
  - Medical Center Klinikum Augsburg, Kinderklinik Augsburg, l. Klinik für Kinder- und Jugendliche, Augsburg
  - Medical Center DRK Kliniken Berlin Westend, Klinik für Kinder- und Jugendmedizin, Berlin
  - Medical Center Evangelisches Klinikum Bethel, Klinik für Kinder- und Jugendmedizin, Bielefeld
  - University Medical Center Ruhr-Universität Bochum, Klinik für Kinder- und Jugendmedizin, Bochum
  - University Medical Center Universitätsklinik Köln, Klinik für Kinder- und Jugendmedizin, Cologne
  - University Medical Center Universitätsklinikum Essen, Kinderklinik I, Neuropädiatrie, Essen
  - University Medical Center Universitätsklinikum Freiburg, Zentrum für Allgemeine Kinder- und Jugendmedizin, Klinik l, Freiburg im Breisgau
  - University Medical Center Universitätsklinikum Gießen und Marburg GmbH, Standort Gießen, Kinderklinik, Abteilung für Kinderneurologie, Sozialpädiatrie u. Epileptologie, Giessen
  - University Medical Center Universitätsmedizin Göttingen, Klinik für Kinder- und Jugendmedizin, Göttingen
  - University Medical Center Universitätsklinikum Hamburg-Eppendorf, Klinik für Kinder- und Jugendmedizin, Hamburg
  - University Medical Center Medizinische Hochschule Hannover, Klinik für Pädiatrische Nieren-, Leber- und Stoffwechselerkrankungen, Hanover
  - University Medical Center Universitätsklinikum des Saarlandes, Homburg, Klinik für Allgemeine Pädiatrie und Neonatologie, Homburg
  - University Medical Center Universitätsklinik Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - University Medical Center Universitätsmedizin Leipzig, Universitätskinderklinik, Leipzig
  - University Medical Center Charité-Universitätsmedizin Berlin, Klinik für Kinder- und Jugendmedizin, Mitte
  - University Medical Center Universitätsklinikum Münster, Klinik für Kinder- und Jugendmedizin, Münster
  - University Medical Center Universitätsmedizin Rostock, Kinder- und Jugendklinik, Rostock

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Boettcher J, Lucke T, Zapf H, Daubmann A, Denecke J, Kersting M, Kalhoff H, Beblo S, Schmidt R, Thiele A, Hohmann S, Kiess W, Muntau AC, Hilbert A, Wiegand-Grefe S. Prevalence of avoidant/restrictive food intake disorder in children and adolescents with rare diseases. Orphanet J Rare Dis. 2026 Jan 31. doi: 10.1186/s13023-026-04233-5. Online ahead of print. PMID 41620754
- [Derived] Boettcher J, Filter B, Denecke J, Hot A, Daubmann A, Zapf A, Wegscheider K, Zeidler J, von der Schulenburg JG, Bullinger M, Rassenhofer M, Schulte-Markwort M, Wiegand-Grefe S. Evaluation of two family-based intervention programs for children affected by rare disease and their families - research network (CARE-FAM-NET): study protocol for a rater-blinded, randomized, controlled, multicenter trial in a 2x2 factorial design. BMC Fam Pract. 2020 Nov 20;21(1):239. doi: 10.1186/s12875-020-01312-9. PMID 33218310